CLINICAL TRIAL: NCT04937322
Title: Radio Frequency Ablation in the Management of Pancreatico-biliary Disorders: A Multicenter Registry.
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 003.GID.2016.D
Record Dates: First submitted 2020-09-21; First posted 2021-06-24 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Bile Duct Cancer; Pancreas Cancer
Keywords: ERCP, endoscopic retrograde cholangiopancreatography; radiofrequency ablation; pancreatico-biliary disorders
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional Endoscopy procedures: All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations for pancreatico-biliary disorders since June 2011 and extending forward through June 2023.
  Interventions: Procedure: Interventional Endoscopy procedures

INTERVENTIONS:
Procedure: Interventional Endoscopy procedures — • All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations and stent insertion(s) for pancreatico-biliary disorders.

SUMMARY:
Bile duct cancer and pancreatic cancer are cancers that cannot be surgically removed. As the cancer grows, it blocks the drainage of the bile ducts that carry digestive juices from the gallbladder and pancreas to the small intestine. ERCP (endoscopic retrograde cholangiopancreatography) is often prescribed during which a tube with a tiny camera attached is inserted through the subject's mouth and advanced to a place in the small intestine where the bile duct empties. Through this scope the doctor enlarges the ducts with tiny balloons and places plastic or metal stents (straws) that help keep the bile ducts open so they can drain properly. However, due to the cancer, the stents are blocked eventually.

The purpose of this registry is to record information and evaluate the impact of endoscopic radiofrequency ablation (RFA) probes in improving the management of bile duct cancer or pancreatic cancer by ablating the tissue in the bile duct(s) before the stent(s) are implanted. By using radiofrequency (RF) energy to heat the tissue in the duct(s) prior to stent(s) insertion, the surrounding tissue becomes coagulated and this may delay tumor growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent implantation(s). The registry will evaluate the efficacy and safety of RFA procedures conducted for pancreatico-biliary disorders

DETAILED DESCRIPTION:
Background

Bile duct cancer and pancreatic cancer are cancers that cannot be surgically removed. As the cancer grows, it blocks the drainage of the bile ducts that carry digestive juices from the gallbladder and pancreas to the small intestine. ERCP (endoscopic retrograde cholangiopancreatography) is often prescribed during which a tube with a tiny camera attached is inserted through the subject's mouth and advanced to a place in the small intestine where the bile duct empties. Through this scope the doctor enlarges the ducts with tiny balloons and places plastic or metal stents (straws) that help keep the bile ducts open so they can drain properly. However, due to the cancer, the stents are blocked eventually.

The purpose of this registry is to record information and evaluate the impact of endoscopic radiofrequency ablation (RFA) probes in improving the management of bile duct cancer or pancreatic cancer by ablating the tissue in the bile duct(s) before the stent(s) are implanted. By using radiofrequency (RF) energy to heat the tissue in the duct(s) prior to stent(s) insertion, the surrounding tissue becomes coagulated and this may delay tumor growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent implantation(s). The registry will evaluate the efficacy and safety of RFA procedures conducted for pancreatico-biliary disorders

Objectives:

The safety and efficacy of various radio frequency ablation probes have been assessed in a series of studies. This multi-center registry has been initiated since June 2011 and is ongoing until June 2017:

* To document the immediate and post procedure clinical performance of radio frequency ablation in a "real world" patient population requiring stent implantation for pancreatico-biliary disorders.
* To assess the immediate and 6 months post procedure adverse event rate in patients.
* To assess the impact of RFA on the life expectancy of patients suffering from pancreatico-biliary malignancies.

Study Design at Coordinating Center - Weill Cornell Medical College Primary site (WCMC):

This study entails review of data from a database protocol [IRB # 1104011642 : collected for non-research related purposes]. The purpose of this protocol is to establish a database that captures all Endoscopic Retrograde Cholangiopancreatography, Endoscopic Ultrasound and Interventional endoscopy cases. Its objective is to assess prospectively the efficacy and safety of these routine procedures to permit identification of technical details about the procedures or other factors, which might be associated with outcome or results. Assessment of these details would help us with problem identification and recommendations to improve health outcomes and quality of life in these patients

The registry will review and document:

* All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations for pancreatico-biliary disorders since June 2011 and extending forward through June 2017.
* Data will be reviewed and collected from database protocol IRB # 1104011642.
* No subject intervention is involved in this study. Subject contact is not needed for database review.

Study Design at Secondary sites:

The registry will review and document:

* All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations for pancreatico-biliary disorders.
* No subject intervention is involved in this study. Subject contact is not needed for retrospective review.
* These sites would have IRB approved protocols to collect and send radio frequency ablation procedure data to the primary site (WCMC). Additionally, the secondary study sites would mention WCMC as an entity that could receive PHI in their prospective protocols and consent/HIPAA forms.
* All secondary study sites' IRB approvals will be sent to the primary/coordinating study center at WCMC. The primary center will then forward these IRB approvals to WCMC IRB as soon as they are received from the secondary study sites.
* Relevant IRB documentation will be maintained at both primary and secondary sites.

Registry Hosting:

The coordinating center and primary site (WCMC) will host the registry on the local servers.

A secure Data management or Electronic Data Capture (EDC) system will be used for data entry, compilation and querying.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations and stent insertion(s) for pancreatico-biliary disorders.
* Above 18 years of age.

Exclusion Criteria:

* Any patient who has not undergone interventional endoscopy with RFA and stent insertion(s).
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have had Interventional Endoscopy procedures done which involved radio frequency ablations and stent insertion(s) for pancreatico-biliary disorders.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Bile Duct Stricture Diameter | June 2011 through June 2021
  Change from Baseline in Bile Duct Stricture Diameter
Adverse Events | June 2011 through June 2021
  Number of Participants with Adverse Events, Type of adverse events, frequency and intensity

SECONDARY OUTCOMES:
survival duration | June 2011 through June 2023
  Documentation of response rates and overall survival duration
stent occlusion-free duration | June 2011 through June 2023
  Documentation of overall stent occlusion-free duration

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
* Data will be collected and entered at/submitted to the primary site (WCMC).
  * A secure Access Database or an alternative secure Electronic Data Capture (EDC) system hosted on the WCMC server will be used for data entry, compilation and reporting.
Supporting Information: Study Protocol, CSR
Time Frame: June 2011 through June 2023